CLINICAL TRIAL: NCT02112669
Title: A Prospective, Multi Center, Study to Evaluate the Safety and Efficacy of the VasQ External Support Device for Brachiocephalic Arteriovenous Fistula
Brief Title: A Multi Center, Study to Evaluate the Safety and Efficacy of the VasQ External Support Device for Arteriovenous Fistulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laminate Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Laminate CD0006
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Vascular Access; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

ARMS (2):
- AV fistula with VasQ (Experimental): Implant VasQ over AV fistula
  Interventions: Device: VasQ
- AV fistula (No Intervention): AV fistula without any adjunct device

INTERVENTIONS:
Device: VasQ
  Arms: AV fistula with VasQ

SUMMARY:
This study is a prospective, multi center, randomized, controlled study of the VasQ in arteriovenous fistulas. The VasQ constraints and directs the geometrical parameters of the fistula as well as the vascular diameter and gradient in the vicinity of the AV shunt. These geometrical constraints direct flow and influence hemodynamics, and hence minimize turbulence and promote laminar flow. The device is designed to improve short term maturation and long term patency of the fistula. The VasQ is a permanent implant intended for use as a subcutaneous arteriovenous conduit support for vascular access.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for creation of a new brachiocephalic fistula who consent to take part in the study.
* Aged > 18
* Male and female participants
* Patients willing and able to attend follow up visits over a period of 6 months

Exclusion Criteria:

* Patients who require revision surgery.
* Having had previous arteriovenous fistula surgery is not a contraindication to recruitment provided the new procedure is not revision surgery
* Target arteries smaller than 3 mm in diameter
* Target vein smaller than 3 mm in diameter
* Stenotic veins on the side of surgery as diagnosed on pre-op ultrasound
* Patients with prior central venous stenosis or obstruction on the side of surgery
* Depth of vein greater than 8 mm (on US) on side of surgery
* Known coagulation disorder
* Prior steal
* Known allergy to nitinol
* Life expectancy less than 6 months
* Inability to give consent and/or comply with the study follow up schedule
* Women of child bearing age

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Primary safety endpoint: Freedom from severe (i.e. performance of daily activities is compromised) or unanticipated device related adverse events | 6 months

SECONDARY OUTCOMES:
Secondary efficacy endpoint: Percentage of AVF physiologically matured | 3 months
  Successful physiological maturation was defined by a minimum of 5 mm cephalic vein diameter with volume outflow greater than 500 mL/min confirmed by color duplex spectral analysis
Secondary efficacy endpoint: Primary patency of the study AVF, defined as percentage of patent AVF free from surgical or endovascular interventions | 6 months
Secondary efficacy endpoint: Cephalic vein outflow as assess with Doppler ultrasound | 1, 3, and 6 months
Secondary efficacy endpoint: Secondary patency of the study AVF, defined as percentage of patent AVF following surgical or endovascular interventions | 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- Sheba Medical Center, Ramat Gan, Israel
- United Kingdom (3):
  - Southmead Hospital, Bristol
  - Guy's Hospital, London
  - St George's Healthcare, London

REFERENCES:
- [Derived] Karydis N, Bevis P, Beckitt T, Silverberg D, Halak M, Calder F. An Implanted Blood Vessel Support Device for Arteriovenous Fistulas: A Randomized Controlled Trial. Am J Kidney Dis. 2020 Jan;75(1):45-53. doi: 10.1053/j.ajkd.2019.05.023. Epub 2019 Aug 22. PMID 31447072